CLINICAL TRIAL: NCT02630836
Title: A Pilot Clinical Trial of ex Vivo Expanded Allogenic Adult Stem Cells Combined With Allogenic Human Bone Tissue (XCEL-MT-OSTEO-BETA) in Proximal Femur Fractures in Elderly Patients
Brief Title: Allogeneic Mesenchymal Stromal Cells in Elderly Patients With Hip Fracture
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Banc de Sang i Teixits (Other)
Collaborators: Fundacion Clinic per a la Recerca Biomédica (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: XCEL-MT-10-03; 2010-024041-78 (EudraCT Number)
Record Dates: First submitted 2015-12-10; First posted 2015-12-15 (Estimated); Last update posted 2017-03-17 (Actual); Status verified 2017-03

CONDITIONS: Femoral Neck Fracture
Keywords: mesenchymal stromal cells; stem cells; elderly; allogeneic; bone marrow; bone regeneration; fracture
MeSH Terms: conditions — Femoral Neck Fractures; Fractures, Bone | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- XCEL-MT-OSTEO-BETA (Experimental): Adult ex-vivo expanded mesenchymal stromal cells from allogeneic bone marrow, cryopreserved, to combine with fibrin glue and cancellous human bone tissue + endomedullary nailing
  Interventions: Drug: XCEL-MT-OSTEO-BETA; Procedure: Surgical treatment
- Standard treatment (Other): Standard surgical treatment with isolated endomedullary nailing
  Interventions: Procedure: Surgical treatment

INTERVENTIONS:
Drug: XCEL-MT-OSTEO-BETA — XCEL-MT-OSTEO-BETA followed by endomedullary nailing
  Arms: XCEL-MT-OSTEO-BETA
Procedure: Surgical treatment — Isolated endomedullary nailing

SUMMARY:
Prospective, unicenter, randomized, open-label, single-dose, two-arms blinded assessor pilot study. Thirty-two (32) elderly patients with hip fracture will be randomized to one of the two treatment-arms (Xcel-MT-osteo-beta or Standard treatment) and be followed for 12 month with the primary objective of safety. Secondary objectives are efficacy through axial tomography and xRay, clinical efficacy and quality of life questionnaire.

DETAILED DESCRIPTION:
Prospective, unicenter, randomized, open-label, single-dose, two-arms blinded assessor phase I-II pilot study.

Thirty-two (32) elderly patients (70-85 years of age) with type 31A2 y 31A3 fracture of the femur (AO/ASIF (Association for the Study of Internal Fixation) classification) admitted at the emergency room of the Hospital Clinic of Barcelona will be randomized 1:1 to one of the two treatment-arms (endomedullary nailing + XCEL-MT-OSTEO-BETA or isolated endomedullary nailing as the standard treatment). Once surgically treated, patients will be followed for 12 month with the primary objective of safety. Secondary objectives are efficacy through axial tomography and xRay, clinical efficacy and quality of life questionnaire (EUROQOL-5D).

ELIGIBILITY:
Inclusion Criteria:

1. Patient between70 and 85 years old
2. Proximal femur fracture type 31A3 31a2 classification AO/ASIF.
3. Deambulation prior to fracture.
4. Written informed consent of the patient or family members.

Exclusion Criteria:

1. Presence of implants at proximal femur level.
2. Presence of local or systemic septic process.
3. Septic arthritis.
4. Dementia of any type.
5. Hematological and biochemical analysis with significant alterations that contraindicate surgery.
6. Patients with positive serology for HIV 1 and 2, Hepatitis B, Hepatitis C and syphilis.
7. Neoplastic disease detected in the last five years or without complete remission.
8. Immunosuppressive status.
9. Patients who received corticosteroids in the 3 months prior to study initiation.
10. Simultaneous participation in another clinical trial or treatment with another investigational product within 3 months prior to inclusion in the study.
11. Other conditions or circumstances that may compromise the patient's participation in the study according to medical criteria.
12. Patient refusal to be followed by a period that may exceed the clinical trial itself.

Ages: 70 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-12; Primary Completion 2017-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
safety of XCEL-MT-OSTEO-BETA in proximal femur fractures by Adverse events, physical exam, laboratory tests. | 12 months
  Adverse events, physical exam, laboratory tests.

SECONDARY OUTCOMES:
efficacy through CT scan | 3 months
  assessment of consolidation by determination of Hounsfield units in CT scan
efficacy through xRay | 1, 3 and 6 months
  assessment of bone callus characteristics by standard radiology
efficacy by clinical assessment | 1, 3 and 6 month
  Clinical assessment by visual analogue scale for pain
efficacy by quality of life questionnaire | 3, 6 and 12 month
  EUROQoL-5D quality of life questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Josep Maria Segur, MD, PhD, Principal Investigator — Hospital Clinic of Barcelona

REFERENCES:
- See also: Blood and Tissue Banc of Catalonia — http://bancsang.net
- See also: Hospital Clínic de Barcelona — http://hospitalclinic.org
- See also: Hospital Clinic Foundation — http://fundacioclinic.org